CLINICAL TRIAL: NCT03816111
Title: A Pragmatic, Registry-based, International, Cluster-randomized Controlled Trial Examining the Use of TEACH-PD Training Modules for Incident PD Patients Versus Existing Practices on the Rate of PD-related Infections
Brief Title: Targeted Education ApproaCH to Improve Peritoneal Dialysis Outcomes Trial
Acronym: TEACH-PD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: The HOME Network (Unknown); Australia and New Zealand Dialysis and Transplant Registry (Unknown); New Zealand Peritoneal Dialysis Registry (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AKTN 17.03
Record Dates: First submitted 2018-12-12; First posted 2019-01-25 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-04

CONDITIONS: Kidney Disease, Chronic; Peritoneal Dialysis Catheter-Associated Peritonitis; Peritoneal Dialysis Catheter Exit Site Infection; Peritoneal Dialysis Catheter Tunnel Infection
Keywords: Training
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEACH-PD Training Curriculum (Experimental): All patients at sites randomized to this arm will receive the TEACH-PD Training Curriculum
  Interventions: Behavioral: TEACH-PD Training Curriculum
- Current Standard PD Training (Active Comparator): All patients at sites randomized to this arm will receive the unit's current PD training materials and plan
  Interventions: Behavioral: Current standard PD training

INTERVENTIONS:
Behavioral: TEACH-PD Training Curriculum — The TEACH-PD training modules have been developed by a core group of renal nurses from the HOME Network in conjunction with senior medical clinicians from the Australasian Kidney Trials Network, eLearning curriculum developers, consumer representatives, and education experts, in line with the International Society for Peritoneal Dialysis guidelines, utilizing modern adult learning principles and best practice eLearning techniques.
  Arms: TEACH-PD Training Curriculum
Behavioral: Current standard PD training — Current PD training materials and plan
  Arms: Current Standard PD Training

SUMMARY:
For many patients peritoneal dialysis (PD) is the preferred form of dialysis to treat kidney disease as it provides greater flexibility and the ability to dialyse at home. However, PD use in Australia has been decreasing over the last 10 years. A big reason for this drop is the risk of infection. The best way to prevent PD related infections is to make sure that patients have good training in PD techniques. The researchers of this study have developed TEACH-PD, a new education package for training both PD nurses and PD patients.

The aim of this study is to find out whether TEACH-PD training reduces the number of PD related infections.

DETAILED DESCRIPTION:
End stage kidney disease is fatal unless treated with dialysis or transplant. Peritoneal dialysis (PD) is a core dialysis modality offering home-based care for patients. PD utilization is frequently threatened beyond 5 years for most patients due to PD-related infections. Patient training is a critical cornerstone of mitigating infection risk and maximizing PD durability (technique survival), but training practices are characterized by a lack of standardization and severe heterogeneity.

There is no high-level evidence to inform PD training. Accordingly, a structured program encompassing how and what to teach PD patients at the inception of PD treatment has the potential to reduce serious PD-related infections, extend the longevity of PD, support cost-effective home-based dialysis care, and reduce costs and health service utilization associated with hospitalization and transition to haemodialysis. TEACH-PD is a standardised modular curriculum for both PD nurse trainers and patients that has been collaboratively developed by renal nurses, doctors, educationalists and patients, aligned to current International Society for Peritoneal Dialysis (ISPD) guidelines, utilizing modern adult learning principles. The TEACH-PD program is feasible and acceptable, as demonstrated in a successful pilot study.

The primary objective of TEACH-PD CRCT (Targeted Education ApproaCH to improve Peritoneal Dialysis outcomes - a Cluster Randomised Controlled Trial) is to determine whether implementation of standardised training modules based on ISPD guidelines targeting both PD trainers and patients results in a longer time to the composite end-point of exit site infections, tunnel infections and peritonitis in incident PD patients compared to existing training practices.

TEACH-PD is a registry-based, pragmatic, multi-center, multinational trial, randomising PD units to implementing TEACH-PD training modules targeted at PD trainers and incident PD patients versus standard existing practices.

An estimated 1,500 patient new to PD will be recruited from at least approximately 42-44 PD units in Australia and New Zealand.The study is being coordinated by the University of Queensland (operating through the Australasian Kidney Trial Network).

The TEACH-PD training modules have been developed by a core group of renal nurses from the HOME Network in conjunction with senior medical clinicians from the Australasian Kidney Trials Network, eLearning curriculum developers, consumer representatives, and education experts, in line with the ISPD guidelines, utilizing modern adult learning principles and best practice eLearning techniques. The modules will be implemented at PD units in Australia and New Zealand to formally evaluate whether, compared with standard care, a standardised training curriculum will reduce the rate of PD-related infections and improve technique survival, resulting in better outcomes for patients receiving PD and significant cost-savings to the community.

ELIGIBILITY:
Inclusion Criteria:

* Patients new to PD;
* Patients > 18 years of age,
* Need to undergo PD training;
* Are able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Time to the first occurrence of any PD-related infection | From the PD start date until first PD-related infection, assessed up to 4 years
  Time to the first occurrence of any PD-related infection including exit site infection, tunnel infection or peritonitis

SECONDARY OUTCOMES:
Time to first exit site infection | From the PD start date until first exit site infection, assessed up to 4 years
  Time to first exit site infection
Time to first tunnel infection | From the PD start date until first tunnel infection, assessed up to 4 years
  Time to first tunnel infection
Time to first episode of peritonitis | From the PD start date until first peritonitis episode, assessed up to 4 years
  Time to first episode of peritonitis
Time to infection-associated catheter removal | From the PD start date until first infection-associated catheter removal, assessed up to 4 years
  Time to infection-associated catheter removal
Incidence of technique failure - 30 days | Assessed at 30 days after transfer to HD or if death occurs within this period
  Incidence of technique failure defined as transfer to haemodialysis for greater than 30-days and/or death within this time
Incidence of technique failure - 180 days | Assessed at 180 days after transfer to HD or if death occurs within this period
  Incidence of technique failure defined as transfer to haemodialysis for greater than 180-days and/or death within this time
Incidence of all-cause hospitalization | Assessed from the PD start date, over up to 4 years
  Incidence of all-cause hospitalization collected via health department hospitalization data linkage
Incidence of all-cause mortality | Assessed from the PD start date, over up to 4 years
  Incidence of all-cause mortality
Participant Quality of Life questionnaire | Completed at baseline, 6, 12, 18 and 24 months
  Participant-reported Quality of Life measured using EQ-5D-5L (EuroQol-5 dimensions questionnaire). EQ-5D-5L measures quality of life using 2 methods - a descriptive scale and a Visual Analogue Scale. The descriptive scale comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/ depression). Each dimension has 5 measurement levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems (5). Numbers associated with levels can be used to report an index score.
  The VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' (100) and 'the worst health you can imagine' (0).
Health-care cost-effectiveness analysis | Assessed from the PD start date, over up to 4 years
  Difference in the incremental cost per Quality Adjusted Life Years gained between treatment arms

OTHER OUTCOMES:
Life participation questionnaire | Completed at baseline and 24 months
  Life participation measured using PROMIS (patient-reported outcomes measurement information system) Short Form - Ability to participate in social roles and activities 6a. PROMIS will measure 6 dimensions (trouble with leisure activities, trouble doing family activities, trouble doing work, trouble doing activities with friends, limiting fun with others and limiting activities with friends). Each dimension has 5 measurement levels: Always (1), Usually, (2), Sometimes (3), Rarely (4) and Never (5).

CONTACTS AND LOCATIONS:
Overall Officials: Neil C Boudville, Prof, Study Chair — University of Western Australia & Sir Charles Gairdner Hospital; Josephine S Chow, Prof, Study Chair — South Western Sydney Local Health District; Yeoungjee Cho, PhD, Study Director — Queensland Health/Princess Alexandra Hospital
Locations (48):
- Australia (33):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Lismore Hospital, Lismore, New South Wales
  - Orange Hospital, Orange, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Nepean/Blacktown Hospital, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Royal Prince Alfred/Concord Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Tamworth Hospital, Tamworth, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Royal Darwin Hospital, Darwin, Northern Territory
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mackay Base Hospital, Mackay, Queensland
  - Logan Hospital, Meadowbrook, Queensland
  - Sunshine Coast University Hospital, Nambour, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital, Launceston, Tasmania
  - Monash Health, Dandenong, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Barwon Health, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- New Zealand (15):
  - Waitakere Hospital, Auckland
  - North Shore Hospital, Auckland
  - Auckland Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Wairau Hospital, Blenheim
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Gisborne Hospital, Gisborne
  - Waikato Hospital, Hamilton
  - Hawke's Bay Hospital, Hastings
  - Nelson Hospital, Nelson
  - Taranaki Hospital, New Plymouth
  - Palmerston North/Whanganui Hospital, Palmerston North
  - Wellington Hospital, Wellington
  - Whangarei Hospital, Whangarei

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication, after deidentification (text, tables, figures and appendices) will be available for individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 2 years and ending 5 years following main publication. Proposals may be submitted up to 5 years following article publication. After 5 years, the data will be available in the investigator's University's data warehouse but without investigator support other than deposited metadata.
Access Criteria: An independent review board will assess proposals based on the following criteria: sound science, benefit-risk balancing and research team expertise.

REFERENCES:
- [Derived] Chow JSF, Boudville N, Cho Y, Palmer S, Pascoe EM, Hawley CM, Reidlinger DM, Hickey LE, Stastny R, Valks A, Vergara L, Movva R, Kiriwandeniya C, Candler H, Mihala G, Buisman B, Equinox KL, Figueiredo AE, Fuge T, Howard K, Howell M, Jaure A, Jose MD, Lee A, Miguel SS, Moodie JA, Nguyen TT, Pinlac G, Reynolds A, Saweirs WWM, Steiner-Lim GZ, TeWhare B, Tomlins M, Upjohn M, Voss D, Walker RC, Wilson J, Johnson DW. Multi-center, pragmatic, cluster-randomized, controlled trial of standardized peritoneal dialysis (PD) training versus usual care on PD-related infections (the TEACH-PD trial): trial protocol. Trials. 2023 Nov 14;24(1):730. doi: 10.1186/s13063-023-07715-0. PMID 37964367